CLINICAL TRIAL: NCT02507726
Title: Multicenter and Open Pilot Clinical Study on the Safety of a New One-piece Convex Appliance in Patients With Enterostomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BBraun Medical SAS (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OPM-G-H-1501
Record Dates: First submitted 2015-07-03; First posted 2015-07-24 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-09

CONDITIONS: Enterostomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Flexima Active Soft convexe (Experimental): Flexima Active soft convexe (1 to 3 appliances per day)
  Interventions: Device: Flexima Active soft convexe

INTERVENTIONS:
Device: Flexima Active soft convexe — The Investigational Device will be used during 14 +- 3 days.

SUMMARY:
This study evaluates the performance of a new 1-piece ostomy convex appliance in patients with enterostomy.

DETAILED DESCRIPTION:
Primary outcome Measure:

To describe Investigational Device performance in term of level of leakage under the skin protector

Secondary Outcome Measure:

* Assessment of the condition of peristomal skin
* Assessment of other performance criteria
* Assessment of AEs for each patient

ELIGIBILITY:
Inclusion Criteria:

* patient is at least 18 years old,
* patient having a colostomy or an ileostomy for at least 1 month,
* patient having a stoma's diameter inferior to 45 mm,
* patient having a flat or flushed or slightly retracted stoma,
* patient using currently a one-piece soft convex or standard ostomy appliance with closed or drainable bags,
* patient using a minimum of 1 product per day with closed pouches or minimum 1 product per two days with drainable pouches
* patient capable to apply and remove the pouch himself or with the help of a caregiver (except health care professional)
* patient having a mental capacity to participate to the study (i.e. to understand the study and to answer to the questions)
* patient agreeing to test investigational product during 14(±3) days.
* patient covered by social security

Exclusion Criteria:

* patient experiencing repeated leakages with his current appliance,
* patient receiving or having received, within the last month, chemotherapy or radiotherapy or corticotherapy,
* patient having a deeply retracted stoma,
* patient currently suffering from peristomal skin complications (bleeding or severe irritation or red and broken skin at the time of inclusion),
* patient already participating in another clinical study or who have previously participated in this investigation,
* pregnant or breast-feeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-06; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Flexima® Active Soft Convex ostomy appliance performance description in term of level of leakage under the skin protector | 14 +- 3 days

SECONDARY OUTCOMES:
Peristomal skin evaluation with DET score scale | baseline and 14 +- 3 days
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | baseline and 14 +- 3 days
Investigational product wear time | 14 +- 3 days
  The patient will complete his patient diary after each Investigational Product removal
Investigational product adhesivity as measured by a Likert scale score (1-4) | 14 +- 3 days
Investigational product flexibility as measured by a Likert scale score (1-4) | 14 +- 3 days
Investigational product conformability as measured by a Likert scale score (1-4) | 14 +- 3 days
Convex ring suppleness of the Investigational product as measured by a Likert scale score (1-4) | 14 +- 3 days
Connection of the Investigational Product belt to the belt hear as measured by a Likert scale score (1-4) | 14 +- 3 days
Residues on the skin after each Investigational Product removal as measured by a Likert scale score (1-4) | 14 +- 3 days
Ease of Investigational Product handling as measured by a Likert scale score (1-4) | 14 +- 3 days
Investigational Product wearing comfort as measured by a Likert scale score (1-4) | 14 +- 3 days
Investigational Product leakage prevention as measured by a Likert scale score (1-4) | 14 +- 3 days
Feeling of Investigational Product security as measured by a Likert scale score (1-4) | 14 +- 3 days
Investigational Product overall satisfaction as measured by a Likert scale score (1-4) | 14 +- 3 days
Use of Investigational Product in the future as measured by a Likert scale score (1-2) | 14 +- 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Patrick RAT, MD, Principal Investigator — University Hospital of Dijon
Locations (1):
- Patrick RAT, Dijon, France